CLINICAL TRIAL: NCT00370474
Title: Multi-Center Assessment of Gain in Navigation Efficiency To Cardiac Resynchronization Therapy
Brief Title: MAGNET CRT Feasibility - Efficiency of LV Lead Placement Comparing Conventional vs. Magnetic Guidance
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Procedure protocol improved - study protocol became obsolete
Sponsor: Stereotaxis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PM-CLIN 001
Record Dates: First submitted 2006-08-29; First posted 2006-08-31 (Estimated); Last update posted 2007-06-18 (Estimated); Status verified 2007-06

CONDITIONS: Cardiac Resynchronization Therapy
Keywords: Bi-V lead; Magnetic Navigation; Cardiac Resynchronization Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Bi-ventricular lead placement

SUMMARY:
Magnetic navigation will permit delivery of the LV lead tip to a prospectively defined location more efficiently and in a higher proportion of patients than is possible with manual navigation.

DETAILED DESCRIPTION:
MAGNET CRT is designed to compare magnetic navigation to manual (i.e., traditional) navigation in placing an over-the-wire (OTW)left ventricle (LV) lead at a target site identified by the investigator. This is a prospective, randomized, multicenter trial in which randomization (2:1, magnetic: manual navigation) will occur after the patient-specific target site is identified on two hardcopy x-ray images of the coronary venogram. The target area will be identified upon review of a venogram of the patient's coronary venous system taken during the current procedure.

Other variables such as navigating through the vasculature to a potential target site (especially if the path is tortuous), achieving good contact with the myocardium, providing repositioning if needed, countering heart motion, retrograde blood flow, and maintaining a stable delivery system during the release of the lead, are all determinants in the success of LV lead placement.

The Magnetic Navigation System (MNS) may thus aid in coronary venous vasculature navigation of guidewires for over-the-wire (OTW) left ventricular (LV) pacing lead placement by assisting in directing the tip of the guidewire, regardless of the tortuosity of a given patient's anatomy.

No investigational products will be used in the conduct of this study. The Niobe® Magnetic Navigation System and all Stereotaxis guidewires and other disposable products to be utilized have received US marketing clearance, and the protocol applications are within their specified intended use.

ELIGIBILITY:
Inclusion Criteria/Exclusion Criteria:

1. The patient is 18 years of age or older.
2. The patient is clinically indicated for left ventricular lead placement as part of a pacing or defibrillator system.
3. The patient may be safely exposed to magnetic fields that exist in Niobe® MNS laboratory.
4. The patient is not participating in any clinical trial or studies that would conflict with the guidewire navigation/LV lead implant protocol for this study.
5. The patient is not pregnant, and if of childbearing potential has completed a pregnancy test which resulted negative.
6. The patient does not have an implanted pacemaker or defibrillator, unless such device will be explanted or otherwise deactivated during this procedure.
7. The patient has no contraindications for contrast dye injection.
8. The patient's diastolic blood pressure is greater than 40 mm Hg.
9. In the opinion of the investigator, the patient's general health status does not preclude participation in the study.
10. In the opinion of the investigator, the patient is a reasonable candidate for participation in this study.
11. The patient is not expected to undergo a heart transplant in the next 6 months.
12. The patient does not have a mechanical triscupid heart valve.
13. The patient has not had a myocardial infarction, unstable angina, percutaneous coronary intervention, or coronary artery bypass graft during the preceding 30 days prior to enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2006-06; Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
The first primary endpoint for this trial is LV lead placement time defined as time from entry of the guidewire into the coronary sinus os to confirmed positioning of the lead tip at the target site
The second primary endpoint will be time from introduction of the LVlead into the introducer sheath to positioning of the lead tip at the target site.

SECONDARY OUTCOMES:
Secondary endpoints include
Skin to Skin time (Time of first skin incision to skin closure)
Success in lead positioning to posterior-lateral location or other identified initial target or other identified initial target determined by 3-month lead-related complication free rate > 80%
Percent of cases with stable lead placement as noted by appropriate sensing and pacing thresholds. by using a pacing system analyzer (PSA)
peri-operatively and pulse generator post-operatively (mean 3-month:
pacing threshold < 2.5 V, amplitude > 3/0 mV, pacing impedance
> 300 Ώ)
Procedural success, defined as the ability to complete the procedure.
CC's of contrast utilized for the procedure.
Total procedure fluoroscopy time.
LV lead placement fluoroscopy time.
Total numbers of guidewires to complete
LV lead placement.
Guidewire-related adverse events.
Procedural adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Ellenbogen, MD, Principal Investigator — Medical Center of Virginia, Richmond, VA
Locations (6):
- United States (6):
  - Northeast Georgia Heart Center, Gainesville, Georgia
  - Central Baptist Hospital, Lexington, Kentucky
  - Caritus St. Elizabeth's Hospital, Boston, Massachusetts
  - Baptist Memphis Hospital, Memphis, Tennessee
  - Trinity Mother Frances, Tyler, Texas
  - Medical Center of Virginia, Richmond, Virginia